CLINICAL TRIAL: NCT05553405
Title: Neuroimmune Mechanisms in Obesity
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No longer able to run study
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Kelly Cosgrove, Professor of Psychiatry and of Neuroscience and of Radiology and Biomedical Imaging, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000031993
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baseline [11C]PBR28 PET Scan (No Intervention): Subjects will complete a 120-minute baseline [11C]PBR28 PET scan.
- Post-Intralipid Infusion [11C]PBR28 PET Scan (Experimental): Subjects will complete a second 120-minute [11C]PBR28 PET scan 4 hours after Intralipid Infusion
  Interventions: Drug: Intralipid Infusion

INTERVENTIONS:
Drug: Intralipid Infusion — Intralipid 20% (a 20% IV fat emulsion) is a sterile, non-pyrogenic fat emulsion prepared for IV administration as a source of calories and essential fatty acids. It is made up of 20% soybean oil, 1.2% egg yolk phospholipids, 2.25% glycerin and water for injection. In addition, sodium hydroxide has been added to adjust the pH so that the final product pH is 8.
  Arms: Post-Intralipid Infusion [11C]PBR28 PET Scan

SUMMARY:
Aim 1: To measure levels of microglia using the radiotracer [11C]PBR28 and PET brain imaging in obese (n=50) vs. lean individuals (n=50). The investigators will recruit 100 subjects who will participate in a single [11C]PBR28 scan to measure levels of TSPO, a marker of microglia.

Aim 2: To determine differences in brain functional connectivity at rest and in response to a decision- making task in obese (n=50) vs. lean individuals (n=50) using fMRI imaging. The same subjects from Aim 1 will participate in a resting state functional magnetic resonance imaging (fMRI) followed by a decision making task during fMRI acquisition.

Aim 3: To assess whether acute elevation of lipid levels through intralipid infusion in lean, healthy individuals (n=20) will induce microglial activation. 20 lean individuals will be recruited to participate in a paradigm that includes a baseline [11C]PBR28 scan, an infusion of intralipid, and a second [11C]PBR28 scan approximately 4 hours post intralipid infusion. The investigators will attempt to utilize subjects from aim 1 in order to use their baseline scans for this paradigm.

Aim 4: To determine whether there are differences in levels of microglia between individuals with and without type 1 diabetes (n=20). 20 patients with diabetes (type 1 diabetes or type 2 diabetes)will be recruited to participate in a single [11C]PBR28 scan to compare to Aim 1 participants.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* Able to read and write English and provide voluntary informed consent
* Physically and psychiatrically healthy by medical history, physical, psychiatric, neurological, EKG and laboratory examinations
* For Aims 1-3: HbA1C < 5.7%
* For Aim 4: HbA1C >6.5% and known diagnosis of T1DM or T2DM

Exclusion Criteria:

* Abnormal labs including Creatinine>1.5mg/dL, Hematocrit < 35% for females and < 39% for males, ALT/AST >2.5X upper limit of normal, abnormal TSH
* Known significant thyroid, hepatic, neurologic, psychiatric, cerebrovascular, or cardiovascular disease
* >5% body weight change in last 6 months
* Current or recent regular steroid use in last 6 months, illicit drug use that is deemed to interfere with results including problematic alcohol use as defined by NIAAA
* Current regular use of psychotropic and/or potentially psychoactive prescription medications
* Regular use of any vitamins/supplements that could affect lipids
* Current regular use of non-steroidal anti-inflammatory medications, statins, or lipid lowering agents
* Vaccination in the last month
* Individuals who are classified as "low binders" for the rs6971 polymorphism (<10% of the population)
* For females, physical or laboratory (-HCG) evidence of pregnancy, seeking pregnancy, or lactating. A urine drug screen and pregnancy test will be performed at screening and prior to the imaging session. Subjects who screen positive will be excluded.

Note: If a subject tests positive for an illicit substance, the PI will determine if the substance would interfere with the results and may terminate participation if applicable. Results of the test would only be noted in the subjects de-identified chart to document the occurrence.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2033-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
Baseline [11C]PBR28 VT values | At baseline
  [11C]PBR28 VT values in our primary regions of interest (PFC and hippocampus) from PET Scan. Linear mixed-effect models will be conducted to evaluate differences in [11C]PBR28 VT values between lean, healthy controls (n=40) and individuals with obesity (n=40), controlling for rs6971 genotype, age, and sex.
Post-Intralipid [11C]PBR28 VT values | Approximately 3 Hours After Intralipid Infusion
  [11C]PBR28 VT values in our primary regions of interest (PFC and hippocampus) from PET Scan. Linear mixed-effect models will be conducted to evaluate differences in [11C]PBR28 VT values between lean, healthy controls (n=40) and individuals with obesity (n=40), controlling for rs6971 genotype, age, and sex.
Baseline Functional Connectivity | At baseline
  ICD values will be obtained from primary a priori regions of interest (vmPFC and hippocampus) with PET Scan. Independent t-tests will be used to compare the ICD data between the study groups.
Post-Intralipid Functional Connectivity | Approximately 3 Hours After Intralipid Infusion
  ICD values will be obtained from primary a priori regions of interest (vmPFC and hippocampus) with PET Scan. Independent t-tests will be used to compare the ICD data between the study groups.
Baseline Microglial Activation | At baseline
  Regional [11C]PBR28 VT values from pre-lipid infusion PET Scan
Post-Intralipid Microglial Activation | Approximately 3 Hours After Intralipid Infusion
  Percent change in regional [11C]PBR28 VT values from pre-lipid infusion PET Scan to post-lipid infusion PET Scan will be calculated across brain regions. Increased microglial activation will be measured as a 20% or more increase in TSPO levels from scan 1 to scan 2

SECONDARY OUTCOMES:
Baseline Visual Attention | At baseline
  Visual attention: response latency to identify card color (log10(ms); higher ~ worse attention).
Post-Intralipid Infusion Visual Attention | Approximately 1 Hour After Intralipid Infusion
  Visual attention: response latency to identify card color (log10(ms); higher ~ worse attention).
Baseline Visual Learning | At baseline
  Visual learning: % of correctly identified repeat cards (arcsine(% correct); higher values ~ better learning).
Post-Intralipid Infusion Visual Learning | Approximately 1 Hour After Intralipid Infusion
  Visual learning: % of correctly identified repeat cards (arcsine(% correct); higher values ~ better learning).
Baseline Verbal Memory | At baseline
  Verbal memory: # of correctly recalled items from a grocery list (3 trials). Verbal recall: # of correctly recalled items from a grocery list after a delay (1 trial; higher ~ better memory/recall).
Post-Intralipid Verbal Memory | Approximately 1 Hour After Intralipid Infusion
  Verbal memory: # of correctly recalled items from a grocery list (3 trials). Verbal recall: # of correctly recalled items from a grocery list after a delay (1 trial; higher ~ better memory/recall).
Baseline Executive Function | At baseline
  Executive function: number of errors navigating a 'hidden' maze (5 trials; higher ~ worse executive function).
Post-Intralipid Executive Function | Approximately 1 Hour After Intralipid Infusion
  Executive function: number of errors navigating a 'hidden' maze (5 trials; higher ~ worse executive function).
Baseline Visual-Motor Processing Speed | At baseline
  Visual-motor processing speed: response latency to detect a card flipped over (log10(ms); higher ~ worse processing speed).
Post-Intralipid Visual-Motor Processing Speed | Approximately 1 Hour After Intralipid Infusion
  Visual-motor processing speed: response latency to detect a card flipped over (log10(ms); higher ~ worse processing speed).
Baseline Working Memory | At baseline
  Working memory: % of correctly identified cards that matched the card presented either one- or two-cards previously (arcsine(% correct); higher ~ better working memory).
Post-Intralipid Working Memory | Approximately 1 Hour After Intralipid Infusion
  Working memory: % of correctly identified cards that matched the card presented either one- or two-cards previously (arcsine(% correct); higher ~ better working memory).
Baseline Social Cognition | At baseline
  Social cognition: response latency to identify the mismatched facial expression based on its emotional content (ms; log10; higher ~ worse social cognition).
Post-Intralipid Social Cognition | Approximately 1 Hour After Intralipid Infusion
  Social cognition: response latency to identify the mismatched facial expression based on its emotional content (ms; log10; higher ~ worse social cognition).
Baseline Reward Responsiveness | At baseline
  Reward responsiveness will be quantified via computerized Probabilistic Reward Task
Post-Intralipid Reward Responsiveness | Approximately 1 Hour After Intralipid Infusion
  Reward responsiveness will be quantified via computerized Probabilistic Reward Task

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Cosgrove, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No